CLINICAL TRIAL: NCT05997966
Title: Investigation of the Effects of Progressive Resistance Exercises on Pain, Functional Activity, Quality of Life and Serum Biomarkers in Individuals With Knee Osteoarthritis
Brief Title: Investigation of the Effects of Progressive Resistance Exercises in Individuals With Knee Osteoarthritis
Acronym: OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meltem Meran Çağlar (Other)
Responsible Party: Sponsor-Investigator, Meltem Meran Çağlar, lecturer, Beykoz University
Organization: Beykoz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeykozU
Record Dates: First submitted 2023-07-22; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee; Exercise Training; Biomarkers
Keywords: Osteoarthritis, Knee; Exercise Training; Pain; Functional Status; Biomarkers; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Exercises Group (Active Comparator): In the exercise group, a home-based exercise program will be applied in addition to a 30-minute walking request twice a week, and will consist of stretching exercises for the lower extremities, isometric exercises and progressive resistance strengthening exercises (IDE) of the hip, knee and ankle. The 12-week home-based IDE program will be applied 2 sets/day for 3 days/week (on non-consecutive days). Resistance bands will be used for resistance in the IDE program. In addition, the exercise intensity in the IDE program will be questioned with the perceived difficulty level (AZD). The AZD scale shows the perceived intensity and pulse rate change during exercise between 6-20. All exercises will be performed without resistance for the first 4 weeks, with AZD levels at 40% of 1 maximum repetition at week 5 to 8, AZD 13-15 (somewhat difficult), and after week 8 to AZD 15-16 (difficult). Progress will be achieved by increasing the number of repetitions.
  Interventions: Other: Progresive Resistance Exercises
- Control Group (Sham Comparator): In the control group, 30 minutes of walking will be requested twice a week, and no other intervention will be made. Individuals in the control group will be called every week by phone for gait follow-up.
  Interventions: Other: No intervation

INTERVENTIONS:
Other: Progresive Resistance Exercises — At the beginning of the study, there will be a home visit (week 0) where the exercises will be taught. Exercise brochures explaining the exercises in written and visual form will also be given to each participant during the first and subsequent home visits. After the first home visit, individuals will be asked to keep an exercise diary prepared by the physiotherapist in order to control the exercises, the occurrence of side effects and dependence on the treatment, and information will be obtained from the individuals by phone calls every week. Two more home visits will take place in weeks 5 and 9 to further the IDE program. Apart from these visits and phone calls, the participant will be allowed to call the physiotherapist if needed. In the exercise group, the 12-week home-based IDE program will be applied 2 sets/day for 3 days/week (on non-consecutive days).
  Arms: Progressive Resistance Exercises Group
Other: No intervation — After a general education about osteoarthritis in the control group, 30 minutes of walking will be requested twice a week, and no other intervention will be made.
  Arms: Control Group

SUMMARY:
It is known that the global socioeconomic burden of individuals with knee osteoarthritis (OA) is on a constantly rising curve. In addition, it is predicted that this burden will increase with the increase in the aging rate of countries. While the evidence level of exercise in the treatment of individuals with knee OA is at A level, a standard exercise program has still not been established for these individuals. One of the most important elements in establishing a standard exercise protocol can be realized by understanding how exercise provides positive effects in these individuals. Today, the gold standard practice used in examining the effectiveness of treatments such as exercise is the follow-up of biomarkers. However, for this purpose, biological fluids (blood, urine, synovial fluid) samples are not taken from individuals with knee OA during routine health controls. Existing laboratory detection methods, especially ELISA analysis, are very detailed, time-consuming and expensive, among the reasons why they cannot be included in routine clinical practice. This situation makes it difficult to examine which biomarkers the exercise programs applied in individuals with knee OA have an effect on and to establish a standard exercise protocol. Therefore, the number of randomized controlled studies examining this issue is very few in the literature, and this number is much less in Turkey. The researchers aimed to create a standard home-based exercise program by examining the effects of the holistic exercise approach for all lower extremity muscles, which the researchers created considering the EMG studies in the literature for individuals with knee OA and the age group to be included in the study, both at the physical (pain, functional status, quality of life) and biochemical level (inflammatory biomarkers that have not been examined together before and whose relationship with OA has been newly discovered).

DETAILED DESCRIPTION:
The researchers aim to evaluate the effectiveness of a home-based holistic progressive resistance exercise program for all lower extremity muscles (hip, knee and ankle circumference) in individuals with knee OA in detail and in a multifaceted manner. In addition, the researchers aim to examine the effect of exercise on serum biomarkers in order to understand whether exercise has an anti-inflammatory effect in these individuals and to establish standard exercise protocols. Thus, when a standard home-based exercise program can be established, it will be ensured that elderly individuals with knee OA, who have problems in reaching health centers, have difficulty in going out due to different health problems, and who are the primary care treatment, will be able to do exercises at home. At the same time, considering the global socioeconomic burden of knee OA, the researchers predict that the home-based exercise program will contribute positively to the country's economy.

All subjects who voluntarily accepted to participate in the study and met the inclusion criteria will be applied four times during the 12-week exercise program (except for the blood draw required for the evaluation of serum biomarker levels). Pain intensity, functional status based on performance and scales, quality of life, lower extremity range of motion, lower extremity muscle strength assessments will be repeated before treatment (0 weeks), 5th and 9th weeks, and after treatment (13th week). These assessments will be made at patients' homes. Blood collection will be done before treatment (week 0) and after treatment (week 13) to examine serum biomarker levels with ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* Having signed the informed consent form,
* Male and postmenopausal female patients aged 50 and over,
* Radiologically and clinically diagnosed with Stage 1 or 2 knee OA,
* Patients with a sedentary life (patients with less than 45 minutes of moderate-intensity activity per week)

Exclusion Criteria:

* Cooperative problem or cognitive impairment,
* BMI > 35 kg/m2,
* Receiving physiotherapy in the last 3 months,
* Steroid injection to the knee joint in the last 6 months,
* Presence of neuromuscular or neurodegenerative disease,
* Presence of cardiorespiratory disease, previous hip, knee, foot-ankle surgeries,
* Use of immunosuppressive drugs,
* Presence of infection or inflammatory disease in any part of the body.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Chair Stand Test | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  A standard chair will be used for the test. First of all, the patient will be asked to sit with his back to the chair. Then, he will be asked to get up from the seat without holding on to the arms of the chair, walk with regular steps at a predetermined length of 3 m, and return to the chair at the end of 3 m. Each patient will be asked to walk at a normal pace and the time will be recorded in seconds with a digital stopwatch.
Timed Up and Go Test | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  A standard chair will be used for the test. First of all, the patient will be asked to sit with his back to the chair. Then, he will be asked to get up from the seat without holding on to the arms of the chair, walk with regular steps at a predetermined length of 3 m, and return to the chair at the end of 3 m. Each patient will be asked to walk at a normal pace and the time will be recorded in seconds with a digital stopwatch. The walking distance will be measured with a tape measure and marked with a colored tape.
Range of Motion | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  Active hip, knee, and ankle joint range of motion will be measured using a universal goniometer. It has been shown that goniometric measurement is a reliable and valid outcome measure in patients with knee OA (Maricar et al., 2016). Hip flexion, abduction, adduction, ankle dorsi and plantar flexion measurements were in supine position; hip extension, knee flexion and extension measurements will be performed in the prone position. Each assessment will be repeated three times, and their average value will be recorded.
Muscle Strength | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  Assessment of muscle strength will be made with a Lafayette manual muscle tester (Lafayette Instrument Company, Lafayette, USA). Measurements will be made in hip abduction, adduction, flexion and extension, knee flexion and extension movements. Measurements will be made in three repetitions for hip abduction, adduction, flexion and extension, with one minute rest between each hip movement and 15 seconds between each repetition. The best values obtained from triple repetitive measurements will be used in the analysis (Mentiplay et al., 2015). Strength measurement of iliopsoas, gluteus maximus, gluteus medius, quadriceps femoris, harmstring, adductor longus and brevis, plantar and dorsi flexor muscles will be performed.
Serum Inflammatory Level | Blood collection will be done before treatment (week 0) and after treatment (week 13) to examine serum biomarker levels with ELISA kits.
  All measurements of serum biomarkers [plasma-soluble TNF-α and TNF-α receptors 1 (sTNFR1), 2 (sTNFR2), serum resistin, IL-1β, IL-6, IL-17, MMP-1 and MMP-3] are strictly aseptic. Under these conditions, 10 ml of venous blood will be drawn from each individual. After centrifugation of the clotted blood at 3000 rpm for 20 minutes, the separated serum samples will be portioned and frozen at -20 C and stored under these conditions until analysis.
Visual Analogue Scale (VAS) | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  It will be used to evaluate the severity of pain. The severity of the pain will be determined by marking a place on a 10 cm straight line drawn between the points of no pain (0) and unbearable pain (10). An increase in the score indicates an increase in pain intensity.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  It is a disease-specific health status measure that is frequently used in patients with knee and hip OA, which consists of three parts (pain, stiffness, and function). WOMAC Turkish version has been shown to be a reliable, valid, sensitive and acceptable outcome measure. WOMAC consists of 24 questions, 5 questions in the pain section, 2 questions in the stiffness section, and 17 questions in the function section. A total score is obtained by scoring each question between 0 and 4 points. Patients are asked to answer the questions by considering the pain, stiffness and activities they have difficulty in performing in the last 24 hours.
Quality of Life Scale-Short Form (SF-12) | Evaluations will be repeated before treatment (week 0), weeks 5 and 9, and post treatment (13 weeks).
  The 12-item short form health questionnaire (SF-12) is a measure that evaluates physical and mental health. It was reported that SF-12, which was created from the original form, SF-36, was easier to apply and had a shorter completion time and was more advantageous to use.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Meran Çağlar, Principal Investigator — Medipol University; bayram ünver, Study Director — Dokuz Eylul University; eda merve kurtuluş, Study Chair — Istanbul Gelisim University; mustafa tekkeşin, Study Chair — istanbul özel sondurak ümran tıp merkezi

IPD SHARING:
Plan to Share IPD: Yes
It is aimed that the data obtained from the research will be published in an academic journal that can be seen and read by everyone, has open access, and is scanned in indexes. It is not aimed to publish in journals that have signed an embargo agreement. Moreover The method part of the academic publication to be produced from the data of our research will be written in detail so that the methods we applied in our research can be repeated by other clinicians or researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study is completed, the data of the study will not be presented in scientific journals and platforms that impose an embargo period that will restrict the sharing of data. Instead, it is aimed to publish scientific publications in high-quality scientific journals and platforms that offer open access.
Access Criteria: It is aimed that the data obtained from the research will be published in an academic journal that can be seen and read by everyone, has open access, and is scanned in indexes. It is not aimed to publish in journals that have signed an embargo agreement. Moreover The method part of the academic publication to be produced from the data of our research will be written in detail so that the methods we applied in our research can be repeated by other clinicians or researchers.